CLINICAL TRIAL: NCT00244647
Title: A Phase 1b, Randomized, Single Blind Study Evaluating RESTEN-MP in Subjects With Focal de Novo Stenosis
Brief Title: A Phase 1b Study Evaluating RESTEN-MP in Subjects With Focal de Novo Stenosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: AVI-4126-CL-06
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease; Coronary Stent Restenosis
Keywords: restenosis; in-stent restenosis
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Drug: RESTEN-MP

SUMMARY:
The process of re-narrowing of a coronary artery following a revascularization procedure such as angioplasty, begins at the time of the procedure. Restenosis has long been considered a major problem for effective long-term interventional success. This often results in repeated procedures to deal with recurrent stenosis (or restenosis) of the original targeted vessel.

There is a substantial body of literature suggesting that local MYC protein production in the injured coronary artery is a major stimulus and potential cause of restenosis that appears after stent placement. This study is based upon the hypothesis that stopping MYC protein production in the vessel has will help reduce restenosis (vessel re-narrowing).

AVI BioPharma Inc., has utilized its proprietary antisense chemistry to design a drug that interferes with MYC production.

This study will evaluate the safety, pharmacokinetics and potential effectiveness of a single intravenous slow-push dose of RESTEN-MP at the time of stent placement to reduce in-stent restenosis following balloon angioplasty and stent placement. The post-dose follow-up period is up to six-months.

DETAILED DESCRIPTION:
The process of restenosis following a revascularization procedure, begins at the time of percutaneous coronary intervention (PCI). Restenosis has long been seen a major impediment of effective long-term interventional cardiology, necessitating repeated procedures to deal with in situ recurrent stenosis of the original targeted vessel. The restenosis rates are between 30 to 50% of patients treated with balloon angioplasty and between 15 to 30% of patients treated with bare metal stents. There is currently high enthusiasm for drug-eluting stents already approved for the market and which have an overall restenosis rate of <3% as reported in published reports for most clinical trial patient populations. However, there are subsets of patients (e.g., diabetic patients and patients with diffuse small vessel disease) that have restenosis rates around 10% despite the use of drug-eluting stents. It is probably too early to conclude that the currently approved drug-eluting stents are a panacea to relieve coronary arterial obstruction due to atherosclerotic heart disease. In fact, with the increased usage of the current drug-eluting stents on the market, there are reports of problems such as late stent malposition, subacute and late thromboses, and aneurysm formations due to the vessel toxicity associated with this method of treatment. There remains a definite need for a simple, safe and durable solution to restenosis.

The development of devices such as intravascular ultrasound has led to a greater understanding of restenosis mechanisms, especially after coronary artery stenting. It is presumed that the pathogenesis of coronary artery restenosis after a revascularization procedure entails two major processes. The first component (viz., recoil and remodeling) involves the mechanical collapse and constriction of the treated vessel; however, coronary stents provide luminal scaffolding that eliminates recoil and remodeling. The second component of coronary artery restenosis after a revascularization procedure is the endothelial response to injury. Whereas, the former focus in modulating the pathophysiological mechanisms involved in restenosis centered mainly on inhibition of platelet aggregation and function, current targets of pharmaceutical agents for this condition have shifted to inhibitors of the cell cycle, smooth muscle cell proliferation and migration, synthesis of extra-cellular matrix, and inflammatory mediators. Many different agents are currently being evaluated in pre-clinical and clinical studies.

AVI-4126, the active ingredient of RESTEN-MP, is a proprietary antisense drug designed to interfere with the ability of human <c-myc> gene to translate mRNA into MYC protein. Slow-push intravenous administration of RESTEN-MP in pharmacological doses in the restenosis porcine model prevented subsequent in-stent stenosis.

In addition to the standard safety assessments, assessments of the potential therapeutic value of RESTEN-MP as a neointimal hyperplasia inhibitor include late loss between the time of stent placement and 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 19 and ≤ 80 years of age.
2. The Subject must be properly consented following FDA regulations and guidelines.
3. Male and Female volunteers with reproductive or childbearing potential must agree to practice adequate birth control methods to protect themselves and partners from conception .
4. Subjects will be scheduled for percutaneous coronary intervention (PCI) due to first time implantation of a Taxus Express stent as a result of stenosis.
5. Subject is an acceptable candidate for coronary artery bypass surgery.
6. The Subject has no more than two lesions within the coronary arterial system requiring stent placement where the diameter of the affected artery or arteries is

   ≥ 2.5 mm and ≤ 4.9 mm based on angiography.
7. The target lesion (and the secondary lesion, if applicable) is ≤ 20 mm in length via angiography.
8. The Subject has had successful placement of a Taxus Express intracoronary stent(s).
9. Subject agrees and is able to return for the scheduled study visits.

Exclusion Criteria:

1. One or more treatable lesions within the coronary arterial system requiring planned or staged intervention prior to the Month One visit.
2. Multi-vessel coronary artery disease involving more than 2 vessels within the coronary arterial system requiring stent placement.
3. Clinically significant findings for any body system that the Principal Investigator determines will exclude a Subject from safely participating in the study.
4. A pregnant or nursing female.
5. Positive history for HIV, HBV or HCV.
6. In-stent restenosis in the target vessel.
7. A target lesion located in an unprotected left main coronary artery or aorto-ostial location or in a bypass graft.
8. Left ventricular ejection fraction < 30%.
9. Angiographic evidence of the target vessel segment angulated ≥ 45º.
10. Angiographic evidence of thrombus or severe calcification in the target lesion.
11. History of bleeding disorders or coagulopathy.
12. NYHA Class III congestive heart failure (CHF).
13. Serum creatinine > 1.5 mg/dL.
14. Clinically active cancer or any medical condition that may lead to study non-compliance or early study termination, confound the results, or is associated with limited life expectancy, i.e., less than 1 year.
15. History of a stroke or trans-ischemic attack (TIA) within 6 months of angioplasty.
16. Unstable ventricular arrhythmias.
17. Evidence of an acute myocardial infarction within 72 hours of the intended treatment (defined as: Q wave or non-Q wave infarction having CK enzymes ≥ 2X the upper laboratory normal with the presence of a CK-MB elevated above the upper limit of normal) or acute myocardial infarction in progress at time of treatment.
18. Known hypersensitivity to aspirin, clopidogrel, or heparin or a contraindication to receive the contrast agent administered during angiographic procedures.
19. Unwilling to accept blood transfusions.
20. Participant in an investigational device or drug study 30 days prior to randomization in this study.
21. A stent other than the Taxus Express is placed.
22. Unsuccessful intracoronary stent placement.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-08

PRIMARY OUTCOMES:
Safety of a single IV slow-push injection of RESTEN-MP administered at the time of Taxus Express™ placement and over a six month surveillance period.

SECONDARY OUTCOMES:
Pharmacokinetics of AVI-4126 when administered as RESTEN-MP.
Evidence of efficacy, based on coronary angiography and IVUS criteria for neointimal hyperplasia and restenosis changes over a 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Porter, M.D., Principal Investigator — University of Nebraska